CLINICAL TRIAL: NCT02118935
Title: Nutritive Effects of Prebiotics on Early Postnatal Behavioral Measures of Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 6023
Record Dates: First submitted 2014-04-04; First posted 2014-04-21 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Behavioral Measures of Tolerance
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Previously marketed cow's milk-based infant formula (Active Comparator)
  Interventions: Other: Previously marketed cow's mlik-based infant formula
- Marketed cow's milk-based infant formula with prebiotics (Experimental)
  Interventions: Other: Marketed cow's milk-based infant formula with prebiotics

INTERVENTIONS:
Other: Previously marketed cow's mlik-based infant formula
  Arms: Previously marketed cow's milk-based infant formula
Other: Marketed cow's milk-based infant formula with prebiotics
  Arms: Marketed cow's milk-based infant formula with prebiotics

SUMMARY:
The study is intended to measure infant comfort, behavior, and sleep when consuming study formula with prebiotics compared to infants who consume a study formula without the prebiotics.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 14-35 days of age at baseline
* Term infant with birth weight of a minimum of 2500 grams
* Solely formula-fed
* Signed Informed Consent and Protected Health Information authorization

Exclusion Criteria:

* History of underlying metabolic or chronic disease, congenital malformation, or immunocompromised
* Feeding difficulties or formula intolerance
* Maternal history of illicit drug use or psychiatric disease

Ages: 14 Days to 35 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Sleep Measures (Amount of time awake and asleep in a 72 hour period) | 14 weeks
Infant State (Infant behavior over a 72 hour period) | 14 weeks

SECONDARY OUTCOMES:
Achieved Weight | 14 weeks
  Total weight gain
Achieved Length | 14 weeks
  Total length gain
Achieved Head Circumference | 14 weeks
  Total head circumference gain
Formula Intake | 14 weeks
Fecal microbiome | Baseline and 112 days of age
Medically-confirmed Adverse Events | 14 weeks
Salivary Cortisol levels | 70 and 120 days of age
Temperament - Infant Behavior Questionnaire | Once at 112 days of age
Sleep Characteristics | 14 weeks
  Amount of waking and sleeping, number of waking and sleep episodes

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lynn Berseth, MD, Study Director — Mead Johnson Nutrition
Locations (7):
- United States (7):
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - Norwich Pediatrics, Norwich, Connecticut
  - Deaconess Clinic, Evansville, Indiana
  - Universty of Kansas Medical Center, Kansas City, Kansas
  - Woburn Pediatrics, Woburn, Massachusetts
  - Pediatric Associates of Mt. Carmel, Cincinnati, Ohio
  - The Jackson Clinic, Jackson, Tennessee